CLINICAL TRIAL: NCT02306330
Title: Assessing Time to Reporting and Clinical Management of Patients With Severe Bacterial and Fungal Infections Between Two Diagnostic Approaches: Matrix-assisted Laser Desorption Ionization-time of Flight Mass Spectrometry Versus Routine Clinical Microbiology for Identifying Pathogens; a Randomized Diagnostic Trial
Brief Title: MALDITOF Versus Routine Clinical Microbiology for Identifying Pathogens; a Randomized Diagnostic Trial
Acronym: MALDITOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government); Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 09HN
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2014-12

CONDITIONS: Bacterial Infections; Fungal Infections
Keywords: Malditof; Malditof MS; matrix-assisted laser desorption ionization-time; identifying pathogens; randomized diagnostic trial
MeSH Terms: conditions — Bacterial Infections; Mycoses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Malditof (Experimental): Specimens of patients (diagnostic aspirates from normally sterile sites: cerebrospinal fluid (CSF), deep abscesses, joint fluid, peritoneal fluid, and pleural fluid, deep tissue biopsies) in Malditof arm will be performed by Malditof instrument to identify the pathogens. It takes 20 minutes for Malditof to identify the pathogens. Then patients will be treated based on these results.
  Interventions: Device: Malditof
- Routine clinical microbiology (Active Comparator): Specimens of patients (diagnostic aspirates from normally sterile sites: cerebrospinal fluid (CSF), deep abscesses, joint fluid, peritoneal fluid, and pleural fluid, deep tissue biopsies) in routine clinical microbiology arm will be conducted by the routine clinical microbiologies and followed the treatment process of the hospital.
  Interventions: Other: Routine clinical microbiology

INTERVENTIONS:
Device: Malditof — Malditof MS system is applied for Malditof group for identifying pathogens. It takes 20 minutes to give the results.
  Arms: Malditof
Other: Routine clinical microbiology — Pathogens will be identified by the routine clinical microbiology of the hospital.
  Arms: Routine clinical microbiology

SUMMARY:
MALDI-TOF MS is capable of directly identifying bacteria and fungi in positive blood cultures, which may be beneficial to patient management. Therefore, MALDI-TOF MS is an important new technology that is becoming routine in developed countries. It is currently unknown whether MALDITOF MS improves diagnostics, costs and patient outcomes in developing countries. This study will assess the clinical impact of a MALDITOF MS system (Maldi Biotyper, Bruker, Germany) in the resource constrained setting of Vietnam and at what cost.

DETAILED DESCRIPTION:
When an eligible specimen from a patient shows pathogen growth, the pathogen identification will be randomized to either MaldiTof or routine diagnostics ('diagnostic pipelines'). Randomization to MaldiTof or routine diagnostics will be 1:1 with stratification by hospital and specimen type (blood vs. other). Isolates grown from all eligible specimens of the same patient will be assigned to the same diagnostic pipeline as the first randomized specimen of that patient.

Allocation to diagnostic arm will be assigned by a web based randomization program. When a pathogen is isolated from a positive eligible specimen, the laboratory technician will log onto the secure randomization program and enter the patient and specimen code. The random diagnostic pipeline allocation will then be generated, informed to the laboratory technician and logged in the study database. In the case of multiple specimens with pathogen growth for a single patient, the unique patient code will trigger the randomization program to generate the same diagnostic arm allocation as the previous sample(s).

ELIGIBILITY:
Inclusion Criteria: Pathogen isolates from the following specimens: blood or diagnostic aspirates from normally sterile sites (including cerebrospinal fluid (CSF), deep abscesses, joint fluid, peritoneal fluid, and pleural fluid, deep tissue biopsies).

Exclusion Criteria:

* Specimens negative for all pathogens
* Specimens from sputum, respiratory or non-surgical wound swabs, nails, mucosal or skin biopsies, urine, fluid from drains, skin swabs and any others not listed in the inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2014-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on optimal antibiotic treatment | Within 24 hours of positive culture (first growth of an eligible specimen).
  Optimal antibiotic treatment is defined as an antibiotic treatment for at least 48 hours since positive culture, targeted to the identified pathogen and later found to cover the organisms antimicrobial resistance profile, while avoiding unnecessary broad spectrum antibiotics (e.g. avoid carbapenems or multiple agents where other agents or single agents would provide sufficient coverage). This study aims to determine The proportion of patients on optimal antibiotic treatment within 24 hours of positive culture (first growth of an eligible specimen).

SECONDARY OUTCOMES:
The total duration of antibiotic treatment | During treatment course, estimated to be 7-10 days.
The total number of antibiotic switches | During treatment course, estimated to be 7-10 days.
Length of ICU stay | During ICU admission, estimated to be 7 days
Length of hospital stay | During hospital admission, estimated to be 12 days
Patient outcome: death, palliative discharge, survived with sequelae, recovered | On or before discharge, estimated to be at 12 days
Costs of microbiological testing | On or before discharge, estimated to be at 12 days
Treatment and hospital costs | On or before discharge, estimated to be at 12 days

OTHER OUTCOMES:
Time from first growth of an eligible specimen to optimal antibiotic treatment. | During hospital admission, estimated to be 0-48 hours
Time from specimen collection of positive eligible specimen to optimal antibiotic treatment | During hospital admission, estimated to be 0-48 hours
The time from first recognition of isolate growth to issue of pathogen identification report | Estimated 0-12 hours
The time from specimen collection to issue of pathogen identification report | Estimated 24-48 hours
Time from first specimen collection to discharge | Estimated to be 12 days
Time from first pathogen identification to discharge | Estimated to be 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Heiman Wertheim, MD, PhD, Principal Investigator — Oxford University of Clinical Research
Locations (2):
- Vietnam (2):
  - National Hospital for Tropical Diseases, Hà Nội
  - Hospital for Tropical Diseases, Ho Chi Minh City

REFERENCES:
- [Derived] Nadjm B, Dat VQ, Campbell JI, Dung VTV, Torre A, Tu NTC, Van NTT, Trinh DT, Lan NPH, Trung NV, Hang NTT, Hoi LT, Baker S, Wolbers M, Chau NVV, Van Kinh N, Thwaites GE, van Doorn HR, Wertheim HFL. A randomised controlled trial of matrix-assisted laser desorption ionization-time of flight mass spectrometry (MALDITOF-MS) versus conventional microbiological methods for identifying pathogens: Impact on optimal antimicrobial therapy of invasive bacterial and fungal infections in Vietnam. J Infect. 2019 Jun;78(6):454-460. doi: 10.1016/j.jinf.2019.03.010. Epub 2019 Mar 23. PMID 30914268
- See also: Oxford University Clinical Research Unit Viet Nam — http://www.oucru.org